CLINICAL TRIAL: NCT04660435
Title: Identification and Monitoring of Resistance to First-line Treatment with CDK 4/6 Inhibitors in Combination with Aromatase Inhibitors in Patients with Metastatic Luminal Breast Cancer Through Non-invasive Biomarkers
Brief Title: To Identify Primary Resistance to CDK4/6 Inhibitors in Breast Cancer
Acronym: TIRESIAS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Sandro Pitigliani (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: Tiresias
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer; ER Positive Breast Cancer; HER2-negative Breast Cancer
Keywords: CDK 4/6 inhibitors; Thymidine Kinase; Palbociclib; Abemaciclib; Ribociclib; circulating tumour DNA; gene expression signatures; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Mandatory: formalin fixed and paraffin embedded (FFPE) tumor block from a baseline biopsy of a metastatic site taken before starting treatment Optional: material from an archival FFPE tumor block from the primary breast tumor Optional: material from one FFPE tumor block of a tissue biopsy from a metastatic site collected upon disease progression to first-line treatment with CDK4/6 inhibitor and AI 24 mL of blood will be collected in EDTA tubes at each time-point Additional 6 ml of whole blood will be collected in EDTA tubes only at baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with ER+/Her2 negative metastatic breast cancer: Patients with ER+/HER2-negative metastatic breast cancer candidate to first-line treatment with a CDK4/6 inhibitor and an aromatase inhibitor as per standard clinical practice
  Interventions: Diagnostic Test: Thymidine kinase activity

INTERVENTIONS:
Diagnostic Test: Thymidine kinase activity — DiviTum® assay determines the enzymatic activity of TK in serum samples
  Other Names: Divitum

SUMMARY:
This is a multi-center biomarkers study aiming to prospectively collect biological samples from patients with ER+ and HER2-negative metastatic breast cancer, who are candidate to first-line treatment with an aromatase inhibitor and a CDK4/6 inhibitor as per standard clinical practice.

Blood and tissue samples will be collected for biomarker analysis, including thymidine kinase1 activity, gene expression signatures and circulating tumor DNA.

DETAILED DESCRIPTION:
Enrolled patients will receive first-line treatment with a CDK4/6 inhibitor + AI (anastrozole, letrozole or exemestane) in accordance with local practice. No drugs will be provided by the study Sponsor. Following disease progression on first-line therapy, subsequent, second-line therapy will be administered at physician discretion and as per physician choice.

For all participating patients, serum and plasma samples will be collected at the following time-points:

* Baseline (< 2 weeks before treatment)
* During treatment with CDK4/6 inhibitors + AI: at day 15 (+/- 2) of the first cycle, day 1 (+/-2) of cycle 2, day 1 (+/- 2) of the cycle closest to the first trial-mandated tumor evaluation (after 12-18 weeks from study inclusion), day 1 (+/- 2) of cycle 6, and every 6 cycles thereafter
* At disease progression or permanent discontinuation of CDK4/6 inhibitors + AI (within 35 days from last CDK4/6 inhibitor dosing)
* During the immediate subsequent treatment (second line) (any type, as per physician choice): at day 1 (+/- 2) of cycle 1 (if > 7 days from last CDK4/6 inhibitors dosing), at day 1 of cycles 3, 6 and every 6 cycles thereafter
* At disease progression or permanent discontinuation of second line treatment (within 35 days from last dosing)

One sample of whole blood will be collected at baseline.

All blood samples will be taken concomitantly with blood draws for routine clinical practice.

To be eligible for the study, availability of material from one formalin fixed and paraffin embedded (FFPE) tumor block from a baseline biopsy of a metastatic site taken before starting treatment is mandatory. Although not mandatory for inclusion, material from an archival FFPE tumor block from the primary breast tumor must also be provided, whenever available. Additionally, material from one FFPE tumor block of a tissue biopsy from a metastatic site collected upon disease progression to first-line treatment with CDK4/6 in and AI will be collected whenever possible

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or older, with a diagnosis of metastatic breast cancer
2. ER-positive and HER2-negative disease as assessed locally either on primary tumor tissue or on a biopsy of a metastasis
3. The patient has not received any prior systemic therapy for metastatic breast cancer (may have received prior hormonal therapy or chemotherapy in the neo/adjuvant setting)
4. The patient is candidate to receive first-line therapy with an aromatase inhibitor (AI) and a CDK4/6 inhibitor per local clinical practice
5. The patient must have evaluable disease according to RECIST 1.1 (either measurable or non-measurable).

   Note: Patients with bone-only disease will be allowed in a specific sub-cohort, which will comprise 10% of the total sample size.
6. Hystologic material from one formalin-fixed, paraffin-embedded (FFPE) tumor block from a diagnostic core or excisional biopsy of a metastatic lesion, taken before study entry must be provided (patients with bone-only disease will be accepted into the trial without a biopsy of the metastatic site). Hystologic material from an additional biopsy (core or excisional) taken at time of disease progression on the study treatment must also be provided, if clinically feasible. When available, hystologic material from an FFPE tumor block from the primary breast cancer must also be submitted.
7. The patient agrees to provide blood samples. at the trial specified time points

Exclusion Criteria:

1. Patients with metastatic disease isolated to the central nervous system (CNS) without metastatic involvement of any other site, unless surgical excision of CNS metastasis has been performed and the tumor tissue is available for the study.
2. Previous or current non-breast malignancies within the last 5 years, with the exception of in situ carcinoma of the cervix and/or adequately treated basal cell or squamous cell carcinoma of the skin

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pre- and post-menopausal patients with luminal (ER-positive and HER2-negative) MBC who have not received prior systemic therapy for MBC, who are candidate to first-line treatment with an aromatase inhibitor and a CDK4/6i as per standard clinical practice.
  Patients must have evaluable disease according to RECIST 1.1 (either measurable or non-measurable). Patients with bone-only disease will be allowed in a specific sub-cohort, which will comprise 10% of the total sample size.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  time from inclusion date to date of first documentation of progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Clinical benefit rate | 5 years
  Complete Response, Partial Response, or Stable Disease ≥24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luca Malorni, Principal Investigator — Azienda USL Toscana Centro - Prato
Locations (1):
- Hospital Santo Stefano, Prato, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malorni L, Tyekucheva S, Hilbers FS, Ignatiadis M, Neven P, Colleoni M, Henry S, Ballestrero A, Bonetti A, Jerusalem G, Papadimitriou K, Bernardo A, Seles E, Duhoux FP, MacPherson IR, Thomson A, Davies DM, Bergqvist M, Migliaccio I, Gebhart G, Zoppoli G, Bliss JM, Benelli M, McCartney A, Kammler R, De Swert H, Ruepp B, Fumagalli D, Maibach R, Cameron D, Loi S, Piccart M, Regan MM; International Breast Cancer Study Group; Breast International Group and PYTHIA Collaborators. Serum thymidine kinase activity in patients with hormone receptor-positive and HER2-negative metastatic breast cancer treated with palbociclib and fulvestrant. Eur J Cancer. 2022 Mar;164:39-51. doi: 10.1016/j.ejca.2021.12.030. Epub 2022 Feb 13. PMID 35172272